CLINICAL TRIAL: NCT02199964
Title: The Effects of Cyclosporin A Emulsion, (Restasis), on the Ocular Surface in Response to Low Humidity Environment in Patients With Dry Eye
Brief Title: The Effects of Cyclosporin A in a Low Humidity Environment, on the Ocular Surface
Acronym: CsA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding was terminated
Sponsor: Baylor College of Medicine (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Steven Pflugfelder, Director of Ocular Surface Clinical Trials, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-33276
Record Dates: First submitted 2014-07-16; First posted 2014-07-25 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Dry Eye
Keywords: Dry eye; environmental stress; artificial tears; cyclosporin; Restasis
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporine; Emulsions; Lubricant Eye Drops; Cyclosporins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cyclosporin 0.05% emulsion (Experimental): used in the eye 4 times a day
  Interventions: Drug: Cyclosporin 0.05% emulsion
- Endura Refresh, Artificial Tears (Active Comparator): Over the Counter artificial tears used in the eye 4 times a day
  Interventions: Drug: Endura, Refresh artificial tears

INTERVENTIONS:
Drug: Cyclosporin 0.05% emulsion — Topical therapy for dry eye
  Other Names: Artificial tears; Cyclosporin 0.05% emulsion (Restasis); Dry Eyes
  Arms: Cyclosporin 0.05% emulsion
Drug: Endura, Refresh artificial tears — Over the counter therapy for dry eye, used 4 times a day
  Other Names: Dry Eyes; Artificial Tears
  Arms: Endura Refresh, Artificial Tears

SUMMARY:
This study will test that hypothesis that topical administration of the FDA approved immunomodulatory agent cyclosporin A emulsion will minimize irritation and ocular surface disease that results from a short term low humidity environmental stress

DETAILED DESCRIPTION:
This is a pilot study designed to evaluate the effect of two conventional dry eye therapies, artificial tears to hydrate and cyclosporine A as an anti-inflammatory, on the irritation symptoms and ocular surface disease of dry eye patients who will be exposed to a low humidity environment for 90 minutes. Patients with dry eye will be enrolled in this study and complete a validated symptom questionnaire and then undergo a complete ocular surface and tear examination to characterize their disease. Enrolled subjects will be exposed to a low humidity environment at the initial evaluation prior to any treatment and will be exposed to a low humidity environment for a second time. They will be randomized to receive either artificial tears or 0.05% cyclosporine A emulsion drop four times a day for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Signature on the written informed consent form
* Patient willingness and ability to return for all visits during the study
* Rapid tear film break up time of seven seconds or less in at least one eye AND
* Both cornea fluorescein staining score greater than or equal to 3 and conjunctival lissamine green staining greater than or equal to 3 in at least one eye
* Ocular Surface Disease Index Symptom Severity score of twenty or greater
* Tear meniscus height less than or equal to 230um
* Intact corneal sensitivity
* Willingness to discontinue use of any current dry eye treatment (except artificial tears) for four weeks prior to enrollment, and during the course of the study

Exclusion Criteria:

* Compromised cognitive ability which may be expected to interfere with study compliance
* Uncontrolled or poorly controlled diabetes or heart or pulmonary disease that could, in the judgment of the investigator, jeopardize subject safety or interfere with the interpretation of the results of the study
* Known hypersensitivity to any components of the artificial tears or cyclosporin A eye drops Anticipated contact lens wear during the study
* History of corneal transplant
* Active ocular infection, uveitis or non-KCS related inflammation
* History of cataract surgery within 3 months prior to enrollment
* History of pterygium removal within 6 months prior to enrollment
* Reduced corneal sensitivity
* Initiation, discontinuation or change in dosage of hormone replacement therapy (HRT), fish oil, evening primrose, flaxseed, or black current seed oil supplements, antihistamines, cholinergic agents, beta-blocking agents, tricyclic or SSRI antidepressants, phenothiazines, or topical or systemic acne rosacea medications in two months prior to enrollment, or anticipated change in dosage during course of study
* Topical ophthalmic medications within prior 4 weeks, or anticipated use of same during the study (except artificial tears)
* Occlusion of the lacrimal puncta either surgically or with temporary collagen punctal plugs within three months prior to study, or anticipated use of same during study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen C. Pflugfelder, MD, Principal Investigator — Baylor College of Medicine, Department of Ophthalmology
Locations (1):
- Alkek Eye Center, Dept of Ophthalmology, Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
The study was terminated early because of loss of funding.

REFERENCES:
- [Background] Alex A, Edwards A, Hays JD, Kerkstra M, Shih A, de Paiva CS, Pflugfelder SC. Factors predicting the ocular surface response to desiccating environmental stress. Invest Ophthalmol Vis Sci. 2013 May 7;54(5):3325-32. doi: 10.1167/iovs.12-11322. PMID 23572103

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment process occurred at the medical clinic of the primary investigator. Recruitment began July 2014 and ended December 2015.
Pre-assignment Details: There were no pre-assignment details.
Period: Overall Study
Arm/Group | Cyclosporin 0.05% Emulsion | Endura Refresh, Artificial Tears
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyclosporin 0.05% Emulsion | Endura Refresh, Artificial Tears | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (9.9) | 58 (4.2) | 54.5 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Corneal Fluorescein Staining
Description: The mean difference in corneal staining using the adjusted CCLR global staining score before and after the environmental challenge at visits baseline and Visit 3/Day 42 when patients were subjected to a 90-minute low humidity stress. Corneal fluorescein staining was graded 0-100 in 5 zones on the cornea. The scores ranged from 0 (minimum) to 500 (maximum). A higher score indicates there was greater cornea disease induced by the low humidity stress on Day 42
Time Frame: 6 weeks
Population: Due to loss of funding, this study was not completed and enrollment ended. Data from only 2 subjects per group was analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cyclosporin 0.05% Emulsion | Endura Refresh, Artificial Tears
Number analyzed (Participants) | 2 | 2
units on a scale | 21.5 (13.44) | 29 (15.6)

2. Secondary Outcome: Eye Irritation Symptoms
Description: The mean difference in subject's scoring of eye irritation symptoms using a VAS (visual analog scale) questionnaire before and after the environmental challenge after treatment at Visit 3/Day 42 when patients were subjected to a 90-minute low humidity stress. Symptoms were graded on a 4 question VAS 0-5 for each question, with scores summed for all questions for a total score that ranges from 0 (minimum) to 20 (maximum) for the pre and post challenge questionnaires. The outcome measure is the difference in the post to pre total score ranging from -20 (maximum improvement) to 20 (maximum worsening). A minus difference indicated the subject had lower irritation symptoms following the lower humidity challenge, while a positive difference indicated the subject had greater irritation following the low humidity challenge on Day 42.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cyclosporin 0.05% Emulsion | Endura Refresh, Artificial Tears
Number analyzed (Participants) | 2 | 2
units on a scale | 1.5 (2.1) | 1 (0)

3. Other Pre Specified Outcome: Conjunctival Goblet Cells
Description: The number of conjunctival goblet cells measured in impression cytology at screening/baseline before and after low humidity exposure at the baseline and Day 42 visits. No (zero) subjects were analyzed because the assay was not performed and data was not collected because the study was terminated due to loss of funding.
Time Frame: 6 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected up to 6 months until study termination.
Description: Adverse event collection was done at each subject visit.
Arm/Group | Cyclosporin 0.05% Emulsion | Endura Refresh, Artificial Tears
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No